CLINICAL TRIAL: NCT05991895
Title: Real-World Study of Iruplinalkib in the Treatment of ALK-Positive Non-Small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Jinming Yu (Other)
Responsible Party: Sponsor-Investigator, Jinming Yu, Director of the hospital, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Other Study IDs: IRU-RWS-001
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Iruplinalkib — Iruplinalkib is administered orally with approximately fixed dosing times each day. The recommended dosage is once daily, on an empty stomach or with food, at 60 mg per dose for the first 1 to 7 days. If tolerated, the dosage is increased to 180 mg per dose starting from the 8th day.

SUMMARY:
This study is a national multicenter real-world investigation aimed at evaluating the real-world effectiveness and safety of Iruplinalkib in the treatment of ALK-positive NSCLC in China.

The study aims to enroll ALK-positive NSCLC patients who have undergone treatment with Iruplinalkib prior to enrollment. Demographic information, medical history, Iruplinalkib-containing treatment regimens, clinical outcomes, adverse events, and related data will be collected for all enrolled patients.

As this study is a real-world investigation, treatment procedures, visit schedules, and examinations will be based on the routine clinical practice of physicians. The primary sources of data for this study will mainly consist of patients' routine medical records or healthcare documentation.

ELIGIBILITY:
Inclusion Criteria:

* Patients willingly contribute their clinical data for this study
* Patients with ALK-positive non-small cell lung cancer
* Age ≥ 18 years
* Patients who have undergone treatment with Iruplinalkib.

Exclusion Criteria:

* Known pregnant or lactating females
* Patients with interstitial lung diseases, drug-related pneumonitis, or radiation pneumonitis require ongoing medical intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALK-positive non-small cell lung cancer
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: JinMing Yu, PhD, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China